CLINICAL TRIAL: NCT04929860
Title: A Cluster Randomised Trial to Evaluate and Intervention to Change Handwashing Behaviour in Rural Indian Households
Brief Title: Intervention to Change Handwashing Behaviour in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WT-001
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2011-06

CONDITIONS: Hygiene; Handwashing; Behaviour
Keywords: diarrhoea; handwashing; hygiene
MeSH Terms: conditions — Behavior; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- handwashing (Active Comparator): This arm receives a scalable social marketing campaign using innovative behaviour change approaches to improve handwashing. The intervention is delivered by a commercial social marketing business unrelated to the investigating organisations
  Interventions: Behavioral: social marketing campaign
- control (No Intervention)

INTERVENTIONS:
Behavioral: social marketing campaign — social marketing campaign delivered over 4 weeks in 4 separate sessions
  Arms: handwashing

SUMMARY:
The research will test the hypothesis that a scalable behaviour change intervention can improve hand-washing practices in rural Indian households. The intervention will be designed using a social marketing approach and will use motivational messages targeting key audiences rather than educational messages about germs and disease which previously have been found ineffective. The intervention will be designed for low-cost, scaleable delivery using a series of visits to target villages by a two-person team on a motorbike. The key goal of the study is to determine the effectiveness of a scaleable, social marketing intervention to promote hand-washing with soap.

The study will take the form of a cluster-randomized, controlled intervention trial. Villages will be randomized to receive either the intervention or no intervention. The primary outcome measure will be the proportion of key events (defecation, faecal contact or food handling) accompanied by hand-washing with soap. These data will be collected by direct observation. A secondary outcome measure will be the number of soap movement episodes. These data will be collected in a sub-sample of households by using electronic motion detectors embedded in bars of soap. Additionally, questionnaires will be used to collect data on social norms, self-reported soap use and habitual soap use. All data will be collected pre and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* households with children of primary school age or younger

Exclusion Criteria:

* households without school-aged or younger children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1747 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Handwashing with soap directly observed | one months after interventions is terminated
  cross sectional survey using direct observation of householders by local study staff

SECONDARY OUTCOMES:
Soap use measured by motion detectors embedded in soap bars | soap movements over one week one month after assessment of the primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- St. John's Research Institute, Palamener, Andhra Pradesh, India